CLINICAL TRIAL: NCT00312962
Title: Neuroscience-Guided Remediation of Cognitive Deficits in Schizophrenia
Brief Title: Effectiveness of Targeted Cognitive Training for Neurological Deficits in People With Schizophrenia
Acronym: CRIS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH068725 (NIH); R01MH068725 (NIH); DATR A2-AISZ
Record Dates: First submitted 2006-04-07; First posted 2006-04-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder; Cognitive Remediation; fMRI
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will use commercially available computer games
  Interventions: Behavioral: Computer games
- 2 (Experimental): Participants will receive targeted cognitive training with neuroplasticity-based software created by Posit Science Corporation
  Interventions: Behavioral: Targeted cognitive training (TCT)

INTERVENTIONS:
Behavioral: Targeted cognitive training (TCT) — TCT includes cognitive remediation exercises that participants practice 1 hour per day, 5 days per week, for 20 weeks. TCT exercises are specifically designed to improve speed and accuracy in the perception of and response to verbal and visuo-spatial targets.
  Arms: 2
Behavioral: Computer games — The control treatment involves commercially available computer games that participants practice 1 hour per day, 5 days per week, for 20 weeks.
  Arms: 1

SUMMARY:
This study will determine the effectiveness of reward-intensive, computer-based targeted cognitive training in improving neurocognitive deficits in people with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a chronic brain disorder that causes severe disability. It is characterized by psychotic symptoms, including hallucinations and delusions. Neurocognitive deficits, such as impaired neurocognitive processing efficiency, also affect people with schizophrenia. This deficiency in the speed and accuracy with which the brain perceives and responds to targets causes scrambled messages to be transmitted in the brain, thereby affecting executive control and memory. Medications are available that effectively treat the psychotic symptoms. The neurocognitive deficits, however, do not subside with medication treatment, and are responsible for the failure to improve the e their psychosocial functioning of people with schizophrenia, even after their psychotic symptoms have gone into remission. The targeted cognitive training (TCT) exercises in this study are specifically designed to improve speed and accuracy in the perception of and response to verbal and visuo-spatial targets. This study will determine the effectiveness of reward-intensive, computer-based TCT in improving neurocognitive deficits in people with schizophrenia.

Participants in this double-blind study will be paired according to IQ and baseline symptom severity. One member of each pair will be randomly assigned to training exercises that use TCT. The other will be assigned to a control intervention, which will involve commercially available computer games. All participants will complete exercises with their assigned intervention for 1 hour per day, 5 days per week, until 90 hours of training has been accumulated. Neuroimaging will be performed on a subgroup of participants to examine changes in brain activation patterns in response to the cognitive training. Upon study completion and at the 6-month follow up visit, participants will be assessed for improvement in the following areas: cognitive performance; symptom profile; quality of life; and social cue recognition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* Good general health
* First language is English
* Clinically stable (i.e., no inpatient hospital stays for 3 months prior to study entry; on stable doses of medication)

Exclusion Criteria:

* History of substance abuse within 6 months prior to study entry
* Neurological disorder
* Any metal in the body, or claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2004-04; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cognitive performance as measured by a neuropsychological battery | Measured at Weeks 8, 14, and 8 and Month 6 follow-up

SECONDARY OUTCOMES:
Symptom profile as measured by clinical interviews | Measured at Weeks 8, 14, and 8 and Month 6 follow-up
Quality of life as measured by clinical interviews | Measured at Weeks 8, 14, and 8 and Month 6 follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Vinogradov, MD, Principal Investigator — UCSF, SFVAMC, NCIRE
Locations (1):
- San Francisco Department of Veterans Affairs Medical Center, San Francisco, California, United States

REFERENCES:
- [Derived] Puig O, Fisher M, Loewy R, Miley K, Ramsay IS, Carter CS, Ragland JD, Niendam T, Vinogradov S. Early- Versus Adult-Onset Schizophrenia as a Predictor of Response to Neuroscience-Informed Cognitive Training. J Clin Psychiatry. 2020 Mar 3;81(2):18m12369. doi: 10.4088/JCP.18m12369. PMID 32141724
- [Derived] Panizzutti R, Hamilton SP, Vinogradov S. Genetic correlate of cognitive training response in schizophrenia. Neuropharmacology. 2013 Jan;64(1):264-7. doi: 10.1016/j.neuropharm.2012.07.048. Epub 2012 Aug 7. PMID 22992330